CLINICAL TRIAL: NCT03343366
Title: Glycemic Control in Type-2 Diabetes Mellitus Patients Through Non-Surgical Periodontal Therapy: A Randomized Controlled Trial
Brief Title: Glycemic Control in T2DM Through Non-Surgical Periodontal Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Collaborators: Higher Education Commission (Pakistan) (Other)
Responsible Party: Principal Investigator, Ambrina Qureshi, Prof. Dr., Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DUHS/DR-O/2017/266
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Chronic Periodontitis; Type 2 Diabetes Mellitus
Keywords: fasting blood glucose; fasting plasma insulin; HOMA-IR insulin resistance; clinical attachment loss
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2 | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: This multi-centric randomized controlled trial (RCT) will be conducted on the baseline sample derived from periodontal clinics of dental institutes of Dow University of Health Sciences. More than 1000 patients will be screened to recruit 150 calculated sample participants (with 50 in each group) with reference to 0.7%, 0.6% reduction and no reduction (0.06%) in the baseline mean HbA1c over a period of 3 months among SRP+AAT, SRP Only and no treatment groups respectively(48) the calculated sample size is 35 in each group (1:1:1) with 99% power of test and 99% confidence interval. Adding 40% dropout rate expected over 6-months follow-up, 49 participants in each group will be required that will be rounded off to 50 in each group (with a ratio of 1:1:1).
Who Masked: Investigator
Masking Description: A parallel group, single blind three-arm design randomized controlled trial (RCT) will be conducted. The examiners, both for periodontal examination and laboratory investigations will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Group 1 (Experimental): The participants in this group will receive a combination of ultrasonic scaling and hand instrumentation required for planing of the root surfaces (SRP) followed by systemic AAT followed by routine warm salt water rinses for 3-5 days and OHI. SRP will be performed using ultrasonic scaling device at medium intensity. In addition to ultrasonic scalar, hand instrumentation (using sharpened and sterilized curettes) may also be used if required to smoothen certain irregular areas of root surface until the surfaces are smooth. Systemic AAT would contain Metronidazole (MET) 400 mg x 3 for 10 days. OHI would include brushing teeth using soft bristles toothbrush and fluoridated toothpaste twice daily (morning after breakfast and night before sleeping) using Modified Bass Technique.
  Interventions: Drug: Metronidazole; Procedure: Scaling Root Planing; Behavioral: Oral Hygiene Instructions
- Test Group 2 (Active Comparator): The participants in this group will receive a combination of Scaling Root Planing followed by routine warm salt water rinses for 3-5 days and OHI. Same procedure for SRP and OHI will be followed as that followed in Test Group 1
  Interventions: Procedure: Scaling Root Planing; Behavioral: Oral Hygiene Instructions
- Control Group 3 (Other): The participants in this group will receive only routine warm salt water rinses for 3-5 days and Oral Hygiene Instructions as that followed in Test Group 1 and Test Group 2. However, after completing six (6) months of evaluation they will be provided DT either in the form of SRP+MET or SRP only in addition to OHI, whichever would be found to have a significant beneficial effect on CP.
  Interventions: Behavioral: Oral Hygiene Instructions

INTERVENTIONS:
Drug: Metronidazole — Systemic AAT would contain Metronidazole (MET) 400 mg x 3 for 10 days
  Other Names: Systemic Adjunct Antibiotic Therapy (AAT)
  Arms: Test Group 1
Procedure: Scaling Root Planing — SRP will be performed using ultrasonic scaling device at medium intensity. In addition to ultrasonic scalar, hand instrumentation (using sharpened and sterilized curettes) may also be used if required to smoothen certain irregular areas of root surface until the surfaces are smooth.
  Other Names: SRP
  Arms: Test Group 1; Test Group 2
Behavioral: Oral Hygiene Instructions — OHI would include brushing teeth using soft bristles toothbrush and fluoridated toothpaste twice daily (morning after breakfast and night before sleeping) using Modified Bass Technique.
  Other Names: OHI

SUMMARY:
It is submitted that incident and prevalent chronic periodontal infection, known as chronic periodontitis (CP) possibly has a causal relationship with diabetes mellitus (DM) having effects on HbA1c, fasting plasma/ blood glucose (FPG/ FBG) and fasting plasma insulin (FPI) levels. Experimental research has suggested that treating CP may improve glycemic control and insulin resistance in Non-Insulin Dependent Type-2 DM patients (T2DM). However, there is limited data concerning the need and effects of adjunct antibiotic therapy (AAT) along with scaling root planning (SRP) in treating CP for long lasting results. Therefore, it is suggested that further research with larger samples must be undertaken for a successful periodontal therapy that may help improve glycemic control at desired levels and longer durations. This study is designed to evaluate effects of periodontal therapy [SRP, metronidazole (MET) and oral hygiene instructions (OHI)] through three-arm trial experiment comprising of SRP+MET+OHI, SRP+OHI and OHI+ Delayed Therapy (DT) groups on HbA1c, FBG, FPI levels and Insulin Resistance calculated through Homeostasis Model Assessment (HOMA-IR) to fill research gap. This study will target large number of individuals (N > 1000) at trial camps known as diabetes-periodontitis (Diab-Per) camps at three different campuses of Dow University of Health Sciences hospitals to be screened for presence of signs and symptoms of chronic periodontitis and type-2 diabetes Mellitus. The selected candidates will be referred to the base camp for further evaluation to be enrolled in trial and recruit 150 participants randomly allocated in each group (50 in each group). Post-therapy follow-up results will be assessed at 1, 3 and 6 months to evaluate short and long term changes in status of CP, FBG, FPI and HbA1c.

DETAILED DESCRIPTION:
The overall evidence that CP has a role in the causal pathway of DM is yet limited and inconsistent. Although intervention research has suggested that treating CP may improve glycemic control and insulin resistance in Type-2 DM patients; yet there is limited data concerning the effects of adjunct antibiotic therapy (AAT) in addition to scaling root planning (SRP) in treating CP for long lasting results. Therefore, it is suggested that further research with bigger samples must be undertaken for a successful periodontal therapy that may help improve glycemic control at desired levels and long durations.

This study is designed to evaluate the effects of periodontal therapy [SRP, metronidazole (MET) and oral hygiene instructions (OHI)] through a three-arm trial comprising of SRP+MET+OHI group, SRP+OHI group and OHI+ Delayed Therapy (DT) group, on HbA1c, FBG, FPI levels and Insulin Resistance calculated through Homeostasis Model Assessment (HOMA-IR) to fill the research gap.

A parallel group, single blind three-arm design randomized controlled trial (RCT) will be conducted over a period of approximately 2 years.

More than 1000 patients will be screened for CP with T2DM to recruit 150 participants for the study. They will be randomly allocated in each group (with 50 in each group). Post-therapy follow-up will be for 1, 3 and 6 months to evaluate short term and long term changes in status of CP, FBG, FPI and HbA1c respectively.

Structured screening form will be used to collect baseline information. HbA1c, FBG levels and IL will be recorded at standardized lab, whereas, CP will be evaluated using standardized periodontal indices by calibrated examiners.

Stata version 11.0 will be used for all kind of data management. Descriptive analysis will be performed using frequency percentages of the categorical variables whereas, mean (standard deviation) will be calculated for all continuous study variables. Inferential statistics will include Chi-square test to assess proportional differences of the categorical variables between the three interventional groups. Whereas, one-way Analysis of Variance test (ANOVA) will be used to evaluate the mean differences of the continuous variables in three different groups. McNemar's Chi-square and Repeated Measure Analysis of Variance (RMANOVA) will be used to assess differences in categorical and continuous variables respectively over time for each intervention group; and particularly to assess second secondary study objective. For insulin resistance HOMA-IR will be calculated to assess an association between CP and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 to 65 years patients suffering from moderate to severe CP at baseline and having HbA1c level ≥7% and <10% at baseline with already diagnosed T2DM at least an year ago will be included as study sample. Moreover, those currently under oral glycemic therapy, having at least 16 natural teeth for the entire study duration and not under any definitive periodontal treatment since last 6 months of baseline visit will be considered as inclusion criteria along with no oral soft tissue lesions and those willing to sign informed consent will be considered to be recruited for this trial

Exclusion Criteria:

* Pregnant or breast feeding women
* Gestational Diabetes
* Patients currently receiving dialysis
* Patients with cardiac pacemakers
* Alcoholic
* Patients with any serious concurrent disease or complication with <1 year of life expectancy.
* Patients suffering from myelo-proliferating disorder (such as sickle cell disease) or under any such treatment that promotes a shift in the hemoglobin pattern.
* Under any anti-inflammatory drugs (daily for >7 consecutive days) within last 2 months of baseline visit, other than low dose aspirin prescribed for Cardio-vascular disease
* Under any systemic immunosuppressive drugs like corticosteroids, cyclosporine etc.
* Under any systemic antibiotics for >7 consecutive days within last four weeks of baseline visit.
* No medication for oral problems during last one month and during follow-up period that may affect interventions and HbA1c levels
* Any change in diabetes related medications in last 3 months of baseline visit, such as change in dose of any one hyperglycemic drug therapy by more than two-fold, addition or subtraction of an oral hypoglycemic agent or addition of insulin.
* Patients requiring any surgical (such as flap-surgery) or any non-surgical periodontal care that is restricted throughout study period depending upon the participants' group he/she may belong to.
* Patients with a history of night-grinding/ bruxism
* Patients with a history of allergic reaction with metronidazole
* Patients with mentally or/ and gross physical disability
* Failure to liaise on with the study protocol over the next 6 months
* With drawl from participation

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Glycated Hemoglobin (HbA1c) | Change from baseline (0) to 3 months and 6 months post intervention
  To examine effects of three non-surgical periodontal therapies through change in HbA1c levels

SECONDARY OUTCOMES:
Clinical Periodontal Measure 1 | Change at 1 and 3 months post intervention in all three groups
  To examine the changes in clinical periodontal measures in terms of Clinical Attachment Loss(CAL)
Clinical Periodontal Measure 2 | Change at 1 and 3 months post intervention in all three groups
  To examine the changes in clinical periodontal measures in terms of Periodontal Pocket Depth (PPD)
Clinical Periodontal Measure 3 | Change at 1 and 3 months post intervention in all three groups
  To examine the changes in clinical periodontal measures in terms of probing (BOP)
Fasting Blood Glucose (FBG) | at 3 and 6 month follow-up between groups.
  To identify an association of clinical periodontal changes on FBG
Fasting Plasma Insulin (FPI) levels | at 3 and 6 month follow-up between groups.
  To identify an association of clinical periodontal changes on FPI
HOMA-IR | at 3 and 6 month follow-up between groups.
  To identify an association of clinical periodontal changes on insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: CHAIRPERSON, DEPARTMENT OF COMMUNITY & PREVENTIVE DENTISTRY, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
It will be available through thesis presentation
Supporting Information: Study Protocol
Time Frame: will be available by mid of year 2020
Access Criteria: it will be accessible only to systematic reviewers on email request only

REFERENCES:
- [Derived] Qureshi A, Haque Z, Bokhari SAH, Baloch AA. Evaluation of HbA1c in type-2 diabetes mellitus patients with periodontitis: preliminary findings of three-arm clinical trial. J Pak Med Assoc. 2020 Aug;70(8):1350-1356. doi: 10.5455/JPMA.22016. PMID 32794485